CLINICAL TRIAL: NCT02920489
Title: Impact of Individualized Timing of Analgesia on the Effectiveness of Labor Analgesia: a Randomized Controlled Trial
Brief Title: Individualized Timing of Analgesia and Effectiveness of Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016[1094]; ChiCTR-IPR-16007976 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2016-07-29; First posted 2016-09-30 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Labor Pain; Analgesia, Obstetrical; Early Medical Intervention
Keywords: severity of labor pain; individualized administration; neuraxial labor analgesia
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Sufentanil; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized epidural analgesia (Experimental): Epidural catheterization will be performed after the beginning of the first stage of labor. Epidural analgesia will begin when asked by parturients and the numeric rating scale of pain is 5 or higher. A loading dose (10 ml mixture of 0.1% ropivacaine and 0.5 ug/ml sufentanil) will be administered through the epidural catheter. After a 20-minute observation, a patient-controlled analgesia pump (containing a mixture of 0.08% ropivacaine and 0.4 ug/ml sufentanil) will be connected to the epidural catheter and programmed to deliver a 6-ml bolus with a 20-minute lockout interval and a 4 ml/h background infusion. Analgesia will be terminated at the end of the third stage of labor.
  Interventions: Drug: Individualized epidural analgesia
- Routine epidural analgesia (Active Comparator): Epidural catheterization will be performed after the beginning of the first stage of labor and the cervix is dilated to 1 cm or more. Epidural analgesia will then begin. A loading dose (10 ml mixture of 0.1% ropivacaine and 0.5 ug/ml sufentanil) will be administered through the epidural catheter. After a 20-minute period observation, a patient-controlled analgesia pump (containing a mixture of 0.08% ropivacaine and 0.4 ug/ml sufentanil) will be connected to the epidural catheter and programmed to deliver a 6-ml bolus with a 20-minute lockout interval and a 4 ml/h background infusion. Analgesia will be terminated at the end of the third stage of labor.
  Interventions: Drug: Routine epidural analgesia

INTERVENTIONS:
Drug: Individualized epidural analgesia — Epidural analgesia will begin when asked by the parturients (during the first stage of labor) and the numeric rating scale is 5 or higher. Analgesia will be terminated at the end of the third stage of labor.
  Other Names: Individualized analgesia with sufentanil and ropivacaine
  Arms: Individualized epidural analgesia
Drug: Routine epidural analgesia — Epidural analgesia will begin when asked by the parturients (during the first stage of labor) and the cervix is dilated to 1 cm or more. Analgesia will be terminated at the end of the third stage of labor.
  Other Names: Routine analgesia with sufentanil and ropivacaine
  Arms: Routine epidural analgesia

SUMMARY:
Neuraxial analgesia is the gold standard to relieve labor pain. A recent "Practice guidelines for obstetric anesthesia" suggests that neuraxial analgesia should be provided in the early stage of labor (cervical dilation < 5 cm) or on a individualized basis. The purpose of this randomized controlled trial is to investigate whether neuraxial labor analgesia administered on an individualized basis can improve analgesia quality and maternal satisfaction.

DETAILED DESCRIPTION:
Neuraxial analgesia is the gold standard to relieve labor pain. It also helps to attenuate maternal anxiety and improve maternal satisfaction. A recent "Practice guidelines for obstetric anesthesia" suggests that neuraxial analgesia should be provided in the early stage of labor (cervical dilation < 5 cm) or, for some special patients, be provided on a individualized basis. Studies showed that, when compared with late administration, early administration of labor analgesia resulted in equivocal findings for spontaneous, instrumented, and cesarean delivery. The investigators hypothesize that neuraxial labor analgesia provided on an individualized basis will further improve analgesia quality and maternal satisfaction. The purpose of this randomized controlled trial is to investigate whether neuraxial labor analgesia administered on an individualized basis can improve analgesia quality and maternal satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparas (aged 18-36 years) with single cephalic term pregnancy;
2. Plan to deliver vaginally, and are considered suitable for a trial of vaginal delivery by obstetricians;
3. Admitted to the delivery room;
4. Agree to receive epidural analgesia during labor.

Exclusion Criteria:

1. History of psychiatric disease (indicate those that are diagnosed before or during pregnancy by psychiatrists);
2. Presence of contraindications to epidural analgesia, which includes: (1) History of infectious disease of the central nervous system (poliomyelitis, cerebrospinal meningitis, encephalitis, etc.); (2) History of spinal or intra-spinal disease (trauma or surgery of spinal column, intra-spinal canal mass, etc.); (3) Systemic infection (sepsis); (4) Skin or soft tissue infection at the site of epidural puncture; (5) Coagulopathy.
3. Other reasons that are considered unsuitable for study participation.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The most severe labor pain score during labor | Assessed at 24 hours after delivery
  Assessed with numeric rating scale, where 0 indicates no pain and 10 the worst pain.

SECONDARY OUTCOMES:
Incidence of instrumental delivery | At the time of delivery
  Incidence of instrumental delivery
Incidence of Cesarean delivery | At the time of delivery
  Incidence of Cesarean delivery
Neonatal Apgar score | At 1 and 5 minutes after delivery
  Neonatal Apgar score
Maternal satisfaction with labor analgesia | Assessed at 24 hours after delivery
  Assessed with the Likert scale, where 1=extremely dissatisfaction, 2=dissatisfaction, 3=neither dissatisfaction nor satisfaction, 4=satisfaction, 5=extremely satisfaction.
Persistent pain score at 24 hours and 42 days after delivery | At 24 hours and 42 days after delivery
  Assessed with numeric rating scale, where 0 indicates no pain and 10 the worst pain.
Rate of breast-feeding | At 24 hours and 42 days after delivery
  Rate of breast-feeding
Incidence of postpartum depression | At 42 days after delivery
  Postpartum depression will be diagnosed as Edinburgh postnatal depression scale of 10 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anim-Somuah M, Smyth RM, Jones L. Epidural versus non-epidural or no analgesia in labour. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD000331. doi: 10.1002/14651858.CD000331.pub3. PMID 22161362
- [Background] Alexander JM, Sharma SK, McIntire DD, Wiley J, Leveno KJ. Intensity of labor pain and cesarean delivery. Anesth Analg. 2001 Jun;92(6):1524-8. doi: 10.1097/00000539-200106000-00034. PMID 11375838
- [Background] Panni MK, Segal S. Local anesthetic requirements are greater in dystocia than in normal labor. Anesthesiology. 2003 Apr;98(4):957-63. doi: 10.1097/00000542-200304000-00024. PMID 12657859
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Sng BL, Leong WL, Zeng Y, Siddiqui FJ, Assam PN, Lim Y, Chan ES, Sia AT. Early versus late initiation of epidural analgesia for labour. Cochrane Database Syst Rev. 2014 Oct 9;2014(10):CD007238. doi: 10.1002/14651858.CD007238.pub2. PMID 25300169
- [Background] Wassen MM, Smits LJ, Scheepers HC, Marcus MA, Van Neer J, Nijhuis JG, Roumen FJ. Routine labour epidural analgesia versus labour analgesia on request: a randomised non-inferiority trial. BJOG. 2015 Feb;122(3):344-50. doi: 10.1111/1471-0528.12854. Epub 2014 May 22. PMID 24849943